CLINICAL TRIAL: NCT07009509
Title: Pilot and Feasibility Testing of a Peer-led Program to Prevent Youth Nicotine Vaping: The YES-CAN! Program
Brief Title: Pilot Study of the YES-CAN! Program to Prevent Youth Nicotine Vaping
Acronym: YES-CAN!
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-1396; 5R34DA058218 (NIH)
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Nicotine Vaping
Keywords: Nicotine Vaping; Adolescents; School; Behavior change; Social norms; Electronic cigarettes
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Intervention Model Description: A credit-earning high school course that includes curriculum related to vaping, health risk communication, and video production will be established and approximately 25-30 10th through 12th grade students will be enrolled. High school students will produce 6-8 short videos intended to increase refusal skills; promote stress management and positive coping; change social norms; prevent vaping initiation; and promote vaping cessation among middle school students. Videos will use a narrative approach and integrate known determinants of vaping. High school students will collaborate with the teacher and researchers to develop discussion guides and skills-building activities based on best practices for substance use prevention. High school students will deliver their videos, along with discussion and supportive activities, to all students in the associated middle school. A text message campaign will reinforce and boost the effectiveness of the classroom sessions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YES-CAN! Intervention (Experimental): A credit-earning middle or high school course that includes curriculum related to vaping, health risk communication, and video production will be established and approximately 25-30 students will be enrolled. Students will produce 6-8 short videos intended to increase refusal skills; promote stress management and positive coping; change social norms; prevent vaping initiation; and promote vaping cessation among middle school students. Videos will use a narrative approach and integrate known determinants of vaping. Students will collaborate with the teacher and researchers to develop discussion guides and skills-building activities based on best practices for substance use prevention. Students will deliver their videos, along with discussion and supportive activities, to all students in the associated middle school. A text message campaign will reinforce and boost the effectiveness of the classroom sessions.
  Interventions: Behavioral: YES-CAN! program

INTERVENTIONS:
Behavioral: YES-CAN! program — Youth Engaged Strategies to Change Adolescent Norms

SUMMARY:
The goal of this pilot study is to determine the feasibility of a randomized trial of the YES-CAN! (Youth Engaged Strategies to Change Adolescent Norms) program to prevent nicotine vaping among adolescents. The program integrates the following evidence-based strategies: youth-adult collaboration; youth-developed narrative videos to convey health messages; peer leaders as change agents; and sustained implementation to change the normative environment. Two middle/high school communities will receive the YES-CAN! intervention. In each school community, a trained teacher will deliver a credit-earning middle or high school class to 25-30 middle or high school students, who will produce 6-8 short videos intended to increase refusal skills; promote stress management and positive coping; change social norms; prevent vaping initiation; and promote vaping cessation among current users. Videos will use a narrative approach and integrate known determinants of vaping. Middle or high school students will collaborate with the teacher and researchers to develop discussion guides and skills-building activities based on best practices for substance use prevention. In 6-8 sessions, middle or high school students will deliver their videos to all students in the associated middle school. A text messaging or other media component will reinforce and boost the effectiveness of the classroom sessions.

Aims for this pilot/feasibility study are:

1. To determine the feasibility and acceptability of implementing the YES-CAN! program
2. To determine the feasibility and acceptability of the research protocols that will be used in a future efficacy trial

DETAILED DESCRIPTION:
This is a pilot/feasibility study of a school-based intervention in which middle and/or high school students develop and deliver a video-narrative-based intervention to middle school students in their school community. To provide evidence of feasibility for the purposes of planning for a large cluster-randomized trial, the investigators will implement the intervention and data collection protocols in two school communities within which students will be followed longitudinally. These school communities are middle schools and/or middle and high school pairs, where each middle school is one of the main schools that feeds into the related high school. The intervention will be delivered over one school year. Baseline and outcome measurements will be conducted via online survey within these schools at baseline, immediately after intervention delivery, and 1-year after baseline.

Within the middle and/or high schools, 25-30 students will participate in the video production and delivery. The school will be encouraged to invite a diverse range of students varying in academic success, gender, socio-economic status, and race/ethnicity to enroll in the credit-earning class. In the fall semester, enrolled students will receive a curriculum related to vaping, health risk communication, and video production. The fall semester will culminate in the completion of 6-8 short narrative videos that are ready for dissemination to middle schools. In the spring semester, students will develop skills and a structure for delivering a vaping prevention program to middle school students. Small groups of participating students will deliver the program in middle school classrooms. Students will be responsible for contacting teachers and scheduling sessions, which will occur mid-February through April, for a total of 6-8 sessions. The middle school sessions will address: health risks of vaping; resistance/refusal skills; healthy ways to cope with stress and anxiety; social skills; and other factors known to be related to nicotine vaping and other forms of substance use in youth. Students will also develop and implement a text message or other type of media campaign for middle school students to boost the effectiveness of the classroom sessions.

Analyses will be conducted using IBM SPSS Statistics 28, SAS Version 9.4 and Mplus Version 8.8. Analyses will be separate for middle school program recipients and the middle/high school program developers. Analyses will address the following domains:

Response rate: An aim is to understand survey response rates and missing data and to develop procedures to address these in the larger trial. Inferential statistics will be used to estimate parameters for key comparisons that assess response rates, student retention/missing data patterns, and random sampling relative to school-level characteristics. The investigators plan to stratify by sex and grade when selecting students for survey participation. This will provide a precise denominator for understanding response rates by these demographics. Response rates will first be assessed descriptively as a proportion of total sampled students within each school, summarized according to age, grade, sex, and race/ethnicity, and compared to overall school-level demographics using t-tests and chi-square or Fisher's exact analyses.

Retention: Given the longitudinal design and student mobility, attrition is anticipated. Students will be invited to complete follow-up surveys even if they missed earlier surveys to allow us to examine missing data patterns. To examine bias generated by attrition over time, the investigators will use independent samples t-tests, chi-square analyses, and regression modeling to compare key baseline variables such as demographic characteristics, vaping behaviors, knowledge, attitudes, perceived norms, and academic aspirations between those who complete 1 and 2 follow-up surveys vs. those lost to follow-up. The investigators will examine attrition in relation to baseline characteristics by regressing baseline constructs (e.g., vaping status, attitudes, norms) on retention status. This regression approach will allow for the testing of interaction terms (e.g., interaction terms of school, grade, and sex with retention status) to determine whether attrition differs by subgroups. Survey response rates will also be compared between middle and high school students and assessed descriptively in terms of time to completion and number of reminders needed. This will provide a way to gauge whether different methods are needed between types of schools, as well as the perceived value of incentives across schools.

Psychometric and distributional evaluation of measures: Baseline demographics and behavioral/attitudinal variables will be summarized using standard descriptive statistics (mean, SD, proportions). Outcome variables are dichotomous, continuous, and ordinal. The investigators will examine the distributional properties of observed data to inform analytic approaches for the larger trial. For psychometric analyses, the investigators will use a split half approach to randomly create EFA and CFA subsamples. Measurement models will be estimated separately for middle school recipient and middle/high school program developer samples, though the investigators will combine the two schools at each level to create the EFA and CFA subsamples (i.e., the middle school and high school EFA/CFA subsamples will include a random selection from each school). The multi-item scales have been derived from prior research, but use of both EFA and CFA will ensure their appropriate use in our local context. Similar constructs (e.g., descriptive norms, injunctive norms) are expected to be related but distinct, though this will be tested empirically using EFA and verified using CFA. EFA modeling will be carried out using maximum likelihood estimation and promax rotation, with final models chosen based on fit (RMSEA), simple structure, and magnitude of factor loadings. The resulting measurement structure from EFA modeling will be estimated in the independent random sample using CFA and interpreted based on model fit (model chi square, RMSEA, and comparative fit index), magnitude and significance of factor loadings, correlations among factors, and internal consistency reliability (Cronbach's alpha).

Subgroup Comparisons: Formal subgroup comparisons (e.g., sex, grade) are proposed to test differences in baseline variables (e.g., vaping use and related attitudes, perceived norms, resistance skills) to better understand how to address unique determinants of vaping among student subgroups in the videos.

School: Analyses will be carried out to compare the two middle schools that receive the program and the two middle/high schools that develop the program on all baseline demographic, behavioral, and attitudinal variables. This is necessary to understand between-school differences for planning a larger trial. Independent samples t-tests and chi-square models, as well as models adjusted for grade and sex using a regression-based framework, may be used. In the larger future efficacy trial, inclusion of additional schools will allow for modeling of school-level fixed and random effects (i.e., three-level model of time nested within students nested within schools).

Sex and Grade: Following the same analytic approach used for school differences, the investigators will test baseline psychosocial variables by sex and grade. The initial approach will be to use bivariate models (t-tests, chi-square) to test sex and grade effects separately, though the investigators will extend this approach to regression modeling of adjusted effects (e.g., sex differences adjusted for grade) as well as potential interaction effects (e.g., sex differences depend on grade).Finally, among middle/high students, the investigators will compare student characteristics measured at baseline between the group of middle/high school students enrolled in the intervention class vs. the broader sample of those students not in the class, both within school and across schools. Student characteristics include sex, age, race/ethnicity, vaping measures (knowledge, attitudes, perceived norms, and behaviors), and positive youth development measures.

ELIGIBILITY:
Inclusion Criteria:

* Children enrolled in middle school grades 6-8 and high school grades 9-12 (age approximately 10-13 and 14-17); adults (over age 18) involved in educational system

Exclusion Criteria:

* Not able to read and write in English or Spanish

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1166 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Ever vaped at baseline | Baseline
  Whether participant has ever vaped, even once or twice. Scores range from "no" (0) to "yes" (1)
Ever vaped at 9 months | 9 months
  Whether participant has ever vaped, even once or twice. Scores range from "no" (0) to "yes" (1)
Every vaped at 12 months | 12 months
  Whether participant has ever vaped, even once or twice. Scores range from "no" (0) to "yes" (1)

SECONDARY OUTCOMES:
Vaping susceptibility at baseline | Baseline
  The average of 2 susceptibility items (I would like to know what vaping feels like; I am curious about vaping) answered on a 5-point scale: 1=completely false, 5=completely true. Scores range from 1 (low susceptibility) to 5 (high susceptibility)
Vaping susceptibility at 9 months | 9 months
  The average of 2 susceptibility items (I would like to know what vaping feels like; I am curious about vaping) answered on a 5-point scale: 1=completely false, 5=completely true. Scores range from 1 (low susceptibility) to 5 (high susceptibility)
Vaping susceptibility at 12 months | 12 months
  The average of 2 susceptibility items (I would like to know what vaping feels like; I am curious about vaping) answered on a 5-point scale: 1=completely false, 5=completely true. Scores range from 1 (low susceptibility) to 5 (high susceptibility)
Days vaped in the past month at baseline | Baseline
  Number of days the participant vaped in the past 30 days, with answers: 0 days (1). 1-2 days (2), 3-5 days (3), 6-9 days (4), 10-19 days (5), 20-29 days (6), all 30 days (7)
Days vaped in past 30 days at 9 months | 9 months
  Number of days the participant vaped in the past 30 days, with answers: 0 days (1). 1-2 days (2), 3-5 days (3), 6-9 days (4), 10-19 days (5), 20-29 days (6), all 30 days (7)
Days vaped in the past 30 days at 12 months | 12 months
  Number of days the participant vaped in the past 30 days, with answers: 0 days (1). 1-2 days (2), 3-5 days (3), 6-9 days (4), 10-19 days (5), 20-29 days (6), all 30 days (7)
Intention to vape at baseline | Baseline
  Participant intention to vape in the next 12 months. Answers include: never (1), once (2), a few times (3), a few times a month (4), a few times a week (5), every day (6).
Intention to vape at 9 months | 9 months
  Participant intention to vape in the next 12 months. Answers include: never (1), once (2), a few times (3), a few times a month (4), a few times a week (5), every day (6).
Intention to vape at 12 months | 12 months
  Participant intention to vape in the next 12 months. Answers include: never (1), once (2), a few times (3), a few times a month (4), a few times a week (5), every day (6).
Vaping knowledge at baseline | Baseline
  A scale that measures knowledge about nicotine vaping. The scale is developed from 7 true/false items. Participant is awarded 1 point for each correct answer. Scores range from 0 (no correct answers) to 7 (all questions answered correctly)
Vaping knowledge at 9 months | 9 months
  A scale that measures knowledge about nicotine vaping. The scale is developed from 7 true/false items. Participant is awarded 1 point for each correct answer. Scores range from 0 (no correct answers) to 7 (all questions answered correctly)
Vaping knowledge at 12 months | 12 months
  A scale that measures knowledge about nicotine vaping. The scale is developed from 7 true/false items. Participant is awarded 1 point for each correct answer. Scores range from 0 (no correct answers) to 7 (all questions answered correctly)
Vaping attitudes at baseline | Baseline
  A scale that measures attitudes towards vaping. The scale is an average of 9 questions measured from completely true (1) to completely false (5). Scale scores range from 1 to 5 with low scores indicating attitudes more favorable towards vaping.
Vaping attitudes at 9 months | 9 months
  A scale that measures attitudes towards vaping. The scale is an average of 9 questions measured from completely true (1) to completely false (5). Scale scores range from 1 to 5 with low scores indicating attitudes more favorable towards vaping.
Vaping attitudes at 12 months | 12 months
  A scale that measures attitudes towards vaping. The scale is an average of 9 questions measured from completely true (1) to completely false (5). Scale scores range from 1 to 5 with low scores indicating attitudes more favorable towards vaping.
Vaping perceived norms at baseline | Baseline
  A scale that measures perceived norms about vaping. The scale is an average of 7 questions measured from completely true (1) to completely false (5). Scale scores range from 1 to 5 with high scores indicating perceived norms supportive of vaping.
Vaping perceived norms at 9 months | 9 months
  A scale that measures perceived norms about vaping. The scale is an average of 7 questions measured from completely true (1) to completely false (5). Scale scores range from 1 to 5 with high scores indicating perceived norms supportive of vaping.
Vaping perceived norms at 12 months | 12 months
  A scale that measures perceived norms about vaping. The scale is an average of 7 questions measured from completely true (1) to completely false (5). Scale scores range from 1 to 5 with high scores indicating perceived norms supportive of vaping.
Vaping resistance skills at baseline | Baseline
  A scale that measures the likelihood of using three strategies for resisting vaping if offered the chance. Items are measured from very likely (1) to very unlikely (5). Scale score is the average of the three items with scores ranging from 1 (very likely to use resistance strategies) to 5 (very unlikely to use resistance strategies).
Vaping resistance skills at 9 months | 9 months
  A scale that measures the likelihood of using three strategies for resisting vaping if offered the chance. Items are measured from very likely (1) to very unlikely (5). Scale score is the average of the three items with scores ranging from 1 (very likely to use resistance strategies) to 5 (very unlikely to use resistance strategies).
Vaping resistance skills at 12 months | 12 months
  A scale that measures the likelihood of using three strategies for resisting vaping if offered the chance. Items are measured from very likely (1) to very unlikely (5). Scale score is the average of the three items with scores ranging from 1 (very likely to use resistance strategies) to 5 (very unlikely to use resistance strategies).
Ever smoked tobacco cigarette at baseline | Baseline
  Whether participant has ever smoked cigarettes, even once or twice Scores range from "no" (0) to "yes" (1)
Ever smoked tobacco cigarette at 9 months | 9 months
  Whether participant has ever smoked cigarettes, even once or twice Scores range from "no" (0) to "yes" (1)
Ever smoked tobacco cigarettes at 12 months | 12 months
  Whether participant has ever smoked cigarettes, even once or twice Scores range from "no" (0) to "yes" (1)

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Crane, PhD, MPH, Principal Investigator — University of Colorado, Denver; Nancy L Asdigian, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Survey data will be fully de-identified, preserved and shared. Scientific data will be made available in CSV format that can be processed in a variety of statistical software packages. To facilitate data use, the study will use standard processing and documentation protocols adopted by the Inter-university Consortium for Political and Social Research (ICPSR) for data formats and dictionaries as well as for variable names, descriptions, and labels. Variable descriptions include a brief explanation of the questionnaire item content or of the constructed measure. Value labels tie individual numeric response codes to descriptive responses from the questionnaire. Public use study data and associated documentation will be made available to the research community free of charge through the Data Sharing for Demographic Research (DSDR) data repository hosted at ICPSR. Datasets in DSDR will be findable and identifiable through a study digital object identifier (DOI) minted by ICPSR.
Supporting Information: Study Protocol
Time Frame: Final submission and release of the study data will occur no later than time of an associated publication or end of the performance period, whichever comes first. Study data deposited in DSDR will be available to the research community in perpetuity. All deidentified study data will be made available as public use data to the research community via DSDR.
Access Criteria: Users of the public use data must register with ICPSR and agree to the Terms of Use, which are designed to protect study participants by limiting data use to scientific research and aggregate statistical reporting, prohibiting attempts to identify study participants, and requiring immediate reporting of any disclosure of study participant identity. Data users also agree not to share or redistribute any data downloads.

REFERENCES:
- [Background] Alzahrani T, Pena I, Temesgen N, Glantz SA. Association Between Electronic Cigarette Use and Myocardial Infarction. Am J Prev Med. 2018 Oct;55(4):455-461. doi: 10.1016/j.amepre.2018.05.004. Epub 2018 Aug 22. PMID 30166079
- [Background] Miech R, Johnston L, O'Malley PM, Bachman JG, Patrick ME. Trends in Adolescent Vaping, 2017-2019. N Engl J Med. 2019 Oct 10;381(15):1490-1491. doi: 10.1056/NEJMc1910739. Epub 2019 Sep 18. No abstract available. PMID 31532955
- [Background] Kechter A, Cho J, Miech RA, Barrington-Trimis JL, Leventhal AM. Nicotine dependence symptoms in U.S. youth who use JUUL E-cigarettes. Drug Alcohol Depend. 2021 Oct 1;227:108941. doi: 10.1016/j.drugalcdep.2021.108941. Epub 2021 Aug 4. PMID 34416679
- [Background] Vogel EA, Prochaska JJ, Ramo DE, Andres J, Rubinstein ML. Adolescents' E-Cigarette Use: Increases in Frequency, Dependence, and Nicotine Exposure Over 12 Months. J Adolesc Health. 2019 Jun;64(6):770-775. doi: 10.1016/j.jadohealth.2019.02.019. PMID 31122507
- [Background] Berry KM, Fetterman JL, Benjamin EJ, Bhatnagar A, Barrington-Trimis JL, Leventhal AM, Stokes A. Association of Electronic Cigarette Use With Subsequent Initiation of Tobacco Cigarettes in US Youths. JAMA Netw Open. 2019 Feb 1;2(2):e187794. doi: 10.1001/jamanetworkopen.2018.7794. PMID 30707232
- [Background] Asdigian NL, Riggs NR, Valverde PA, Crane LA. Reducing Youth Vaping: A Pilot Test of the Peer-Led "Youth Engaged Strategies for Changing Adolescent Norms!" (YES-CAN!) Program. Health Promot Pract. 2023 Sep;24(5):956-962. doi: 10.1177/15248399221100793. Epub 2022 Jun 9. PMID 35678642
- [Background] Tobacco prevention tool kit. Stanford Medicine Tobacco Prevention Tool Kit website. https://med.stanford.edu/tobaccopreventiontoolkit.html. Accessed January 7, 2023.
- [Background] National Youth Tobacco Survey. https://www.cdc.gov/tobacco/data_statistics/surveys/nyts/index.htm. 2022. Accessed March 5, 2023.
- [Background] Monitoring the Future Survey. https://nida.nih.gov/research-topics/trends-statistics/monitoring-future. 2021. Accessed March 5, 2023.
- [Background] Youth Risk Behavior Survey. https://www.cdc.gov/healthyyouth/data/yrbs/index.htm 2020. Accessed March 5, 2023.
- [Background] Population Assessment of Tobacco and Health Study (PATH, youth interview). https://pathstudyinfo.nih.gov/. 2022. Accessed March 5, 2023.
- [Background] Gorukanti A, Delucchi K, Ling P, Fisher-Travis R, Halpern-Felsher B. Adolescents' attitudes towards e-cigarette ingredients, safety, addictive properties, social norms, and regulation. Prev Med. 2017 Jan;94:65-71. doi: 10.1016/j.ypmed.2016.10.019. Epub 2016 Oct 20. PMID 27773711
- [Background] Farrelly MC, Duke JC, Crankshaw EC, Eggers ME, Lee YO, Nonnemaker JM, Kim AE, Porter L. A Randomized Trial of the Effect of E-cigarette TV Advertisements on Intentions to Use E-cigarettes. Am J Prev Med. 2015 Nov;49(5):686-693. doi: 10.1016/j.amepre.2015.05.010. Epub 2015 Jul 7. PMID 26163170
- [Background] Spoth R, Guyll M, Trudeau L, Goldberg-Lillehoj C. Two studies of proximal outcomes and implementation quality of universal preventive interventions in a community-university collaboration context. J Community Psychol. 2002;30(5), 499-518. https://doi.org/10.1002/jcop.10021
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Peterson NA, Lowe JB, Hughey J, Reid RJ, Zimmerman MA, Speer PW. Measuring the intrapersonal component of psychological empowerment: confirmatory factor analysis of the sociopolitical control scale. Am J Community Psychol. 2006 Dec;38(3-4):287-97. doi: 10.1007/s10464-006-9070-3. PMID 16977501
- [Background] Ozer EJ, Schotland M. Psychological empowerment among urban youth: measure development and relationship to psychosocial functioning. Health Educ Behav. 2011 Aug;38(4):348-56. doi: 10.1177/1090198110373734. Epub 2011 May 23. PMID 21606379
- [Background] Melchior A. Center for youth and communities: Earth Force evaluation instrument. Unpublished document. 2011.
- [Background] Furlong MJ, O'Brennan LM, You S. Psychometric properties of the ADD HEALTH school connectedness scale for 18 sociocultural groups. Psychol Schools. 2011;48(10):986-997. https://doi.org/10.1002/pits.20609
- [Background] Greene K, Yanovitzky I, Carpenter A, Banerjee SC, Magsamen-Conrad K, Hecht ML, Elek E. A Theory-Grounded Measure of Adolescents' Response to a Media Literacy Intervention. J Media Lit Educ. 2015;7(2):35-49. PMID 28042522
- [Background] IBM Corp. Released 2021. IBM SPSS Statistics for Windows, Version 28.0. Armonk, NY: IBM Corp.
- [Background] SAS/STAT software, v. 9.4 of the SAS System for Windows. Copyright © 2014 SAS Institute Inc. Cary, NC, USA.
- [Background] Muthén LK, Muthén BO. (1998-2017). Mplus User's Guide. Eighth Edition. Los Angeles, CA: Muthén & Muthén.